CLINICAL TRIAL: NCT04322747
Title: Hearing Changes After Skull Base and Mastoid Surgery
Brief Title: Hearing Changes After Surgery
Status: Withdrawn | Type: Observational
Why Stopped: COVID protocols caused extreme delays.
Sponsor: Gateway Biotechnology, Inc. (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 19090236; 3R41DC017406-01S1 (NIH)
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hearing Loss
Keywords: Hearing changes; Non-surgical ear; Hearing loss; Vibration exposure; Skull-based surgery; Un-operated ear
MeSH Terms: conditions — Hearing Loss | interventions — Acoustic Impedance Tests; Audiometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants scheduled to undergo skull-based surgery: Participants scheduled to undergo skull-based or mastoid surgery as part of their standard care will receive Audiometry for extended high frequencies, DPOAE, ECochG before and after the procedure in the non operated ear.
  Interventions: Diagnostic Test: Distortion product otoacoustic emissions (DPOAE)

INTERVENTIONS:
Diagnostic Test: Distortion product otoacoustic emissions (DPOAE) — Audiometry for extended high frequencies, DPOAE, and, ECochG measurements will be collected before and after skull-based surgeries.
  Other Names: Electrocochleaography/Electrophysiological testing; Tympanometry; Audiometry

SUMMARY:
The purpose of this study is to measure the potential effects of surgical drilling noise and/or vibration exposure on the hearing in the ear contralateral to the surgical site during skull-based surgeries

DETAILED DESCRIPTION:
High-speed drills that are capable of producing elevated levels are used during skull based surgeries (Hilmi et al., 2011; Yu et al., 2014). Recently, it has been shown that surgical drilling may have a temporary effect on the amplitude of the otoacoustic emissions of the ear contralateral to the surgical site (Baradaranfar et al., 2015; Shenoy et al., 2015), however the temporary effects of surgical noise or vibration on the hearing of the non-surgical related ear needs to be better quantified. This study aims to to measure the potential effects of surgical drilling noise and/or vibration exposure on the hearing in the non operative ear, during surgical site during skull-based or mastoid surgeries. As part of the study patient will receive Audiometry for extended high frequencies, DPOAE, ECochG before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* participants are undergoing a skull-based or mastoid surgery for treatment of an affected ear
* participants have normal or near-normal hearing thresholds in the un-operated ear

Exclusion Criteria:

* participants have hearing loss (PTA > 40 dB HL) in pure tone audiometry testing before surgery in the un-operated ear
* participants have medical conditions after the surgery which prevents having hearing tests
* participants have abnormal tympanometric results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to undergo skull-based and mastoid surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Difference of 5 dB or more between Pre- and Post-surgery DPOAE Measurements at any Frequency | pre-surgery, immediately after surgery, up to one month after surgery
  DPOAE measurement using Interacoustics Titan DPOAE440 measurement tool is 5dB or greater from pre-surgery measurement to post-surgery measurement
Number of Participants with No change between Pre- and Post-surgery DPOAE Measurements | pre-surgery, immediately after surgery
  DPOAE measurement using interacoustics titan measurement tool has not changed or is less than 5dB from pre-surgery measurement to post-surgery measurement

CONTACTS AND LOCATIONS:
Overall Officials: Partha Thirumala, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Baradaranfar MH, Shahbazian H, Behniafard N, Atighechi S, Dadgarnia MH, Mirvakili A, Mollasadeghi A, Baradaranfar A. The effect of drill-generated noise in the contralateral healthy ear following mastoid surgery: The emphasis on hearing threshold recovery time. Noise Health. 2015 Jul-Aug;17(77):209-15. doi: 10.4103/1463-1741.160691. PMID 26168951